CLINICAL TRIAL: NCT02525289
Title: Study of Impact of Three Body Positioning Strategies in the Drainage Fluids in the Immediate Postoperative Period in Patients After Coronary Artery Bypass Surgery
Brief Title: Impact of Three Body Positioning Strategies in the Drainage Fluids After Coronary Artery Bypass Surgery
Acronym: positioning
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Emilia Nozawa, PT PhD, principal investigator, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 141372
Record Dates: First submitted 2015-07-20; First posted 2015-08-17 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Coronary Artery Disease
Keywords: mobility; coronary artery bypass; positioning; body
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control Group (No Intervention): six hours after extubation receiving breathing exercises. After 48 hour postoperative time, sitting on armchair and keeping the erect position and walking in the same place.
- Bed Rotation Group (Active Comparator): six hours after extubation receiving breathing exercises and submitted the continuous rotational bed therapy in the first postoperative day until 48 hours.
  Interventions: Other: Bed Rotation Group
- Orthostatic Group (Active Comparator): six hours after extubation receiving breathing exercises and changing the body position following the sequence: sitting on the bed, sitting on the bed with the feet on the floor , standing and walking in the same place, in the first postoperative day until 48 hours.
  Interventions: Other: Orthostatic Group

INTERVENTIONS:
Other: Bed Rotation Group — Patients received continuous lateral rotation by a mechanical device (Hill Rom Bed Rotation), consecutive cycles of to left and right side, plus supine position during 30 seconds for pause, in the first postoperative day until 48 hours. Additional breathing exercises.
  Arms: Bed Rotation Group
Other: Orthostatic Group — Patients were seated on the bed 6 hours post extubation for two hours. After, sitting in the bed with their feet on the floor for two minutes; standing up and walking in the place for two minutes, in the first 24 hours and 48 hours postoperative. Additional breathing exercises.
  Arms: Orthostatic Group

SUMMARY:
To investigate different strategies of body positioning associated to early corporal mobilization and verify the impact int the time and quantification of thoracic and mediastinal drainage, pulmonary complications and time of intensive care units in hospitals stay. After first six hours post extubation in the first postoperative day and after evaluation and inclusion in the study, patients were randomized in three groups for receiving different strategies of body positioning associated to early mobilization with help of bed Hill Rom (Hill Rom Batesville@): Group 1: Control (GC n=33); Group 2: Continuous Lateral Rotation Group (TRCL n=34); Group 3:Positioning in sitting and Orthostatic (ORT n=34).

DETAILED DESCRIPTION:
Coronary artery bypass surgery can lead to pulmonary complications like pleural effusion and pneumonia. These complications increase the length of stay and the immobility time. The investigators aim was to assess the impact of early mobilization of fluids drainage of chest tubes and the incidence of pulmonary complications. A prospective, randomized study included 101 patients divided in three groups. In the Control Group (CG:n=33) the patients were seated in armchair in the first 48 hours postoperative time. The Group (TRCL n=34) a Continuous Rotational Bed Therapy was instituted six hours post extubation in the first 24 hours and it comprised with by consecutive cycles of lateral rotation to the left and right side, and supine position with 30 seconds for pauses (using a Hill Rom Rotational Bed Device) witch stopped when need to perform routine measurements the hemodynamics measurements and clinical controls by nursing crew.The group ( ORT n=33) following the sequential steps T1: sitting in the bed for 2 hours, T2: sitting on the bed with their feet on the floor for 2 minutes and T3: the patients stoos up and walked on the spot for 2 minutes. Hemodynamics and oxygenation measurement before and after each intervention.

ELIGIBILITY:
Inclusion Criteria:

* first postoperative day of cardiovascular surgery 6 hours after extubation
* EFVE> 35%
* writen inform consent

Exclusion Criteria:

* neurological alteration
* hemodynamics instability with PAM < 60 mmHg
* blood
* pneumothorax or broncopleural
* arritymias

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2012-11; Primary Completion 2013-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
volume of drainage fluids | 48 hours
  measure of volume of drainage fluids (mililiter) pre and post intervention until extract the mediastinal and/or thoracic tube

SECONDARY OUTCOMES:
score of pulmonary complications | 7 days
  incidence of postoperative pulmonary complications, was scored by a blinded independent investigator on an ordinal scale of 1 to 4

CONTACTS AND LOCATIONS:
Overall Officials: Filomena G Gallas, PHD, Study Director — University of Sao Paulo; Ludhmila A Hajjar, PHD, Study Chair — University of Sao Paulo Medical School; Maria Ignêz Z Feltrim, PHD, Study Director — Heart Intsitute (InCor) Hospital das Clinicas - FMUSP; Camila CM Buzzeto, PT, Study Chair — Heart Institute (InCor) Hospital das Clinicas - FMUSP; Vera RM Coimbra, PT, Study Chair — Heart Institute (InCor) Hospital das Clinicas _ FMUSP; Adriano RB Rodrigues, Nursing, Study Chair — Heart Intitute (InCor) Hospital das Clinicas _ FMUSP; Cristiane D Gonçalves, PT, Study Chair — Heart Intitute (InCor) Hospital das Clinicas _ FMUSP

REFERENCES:
- [Result] Kirkeby-Garstad I, Stenseth R, Sellevold OF. Post-operative myocardial dysfunction does not affect the physiological response to early mobilization after coronary artery bypass grafting. Acta Anaesthesiol Scand. 2005 Oct;49(9):1241-7. doi: 10.1111/j.1399-6576.2005.00854.x. PMID 16146459
- [Result] Goldhill DR, Imhoff M, McLean B, Waldmann C. Rotational bed therapy to prevent and treat respiratory complications: a review and meta-analysis. Am J Crit Care. 2007 Jan;16(1):50-61; quiz 62. PMID 17192526
- [Result] Hulzebos EH, Helders PJ, Favie NJ, De Bie RA, Brutel de la Riviere A, Van Meeteren NL. Preoperative intensive inspiratory muscle training to prevent postoperative pulmonary complications in high-risk patients undergoing CABG surgery: a randomized clinical trial. JAMA. 2006 Oct 18;296(15):1851-7. doi: 10.1001/jama.296.15.1851. PMID 17047215
- [Result] Morris PE, Goad A, Thompson C, Taylor K, Harry B, Passmore L, Ross A, Anderson L, Baker S, Sanchez M, Penley L, Howard A, Dixon L, Leach S, Small R, Hite RD, Haponik E. Early intensive care unit mobility therapy in the treatment of acute respiratory failure. Crit Care Med. 2008 Aug;36(8):2238-43. doi: 10.1097/CCM.0b013e318180b90e. PMID 18596631
- [Result] Perme C, Chandrashekar R. Early mobility and walking program for patients in intensive care units: creating a standard of care. Am J Crit Care. 2009 May;18(3):212-21. doi: 10.4037/ajcc2009598. Epub 2009 Feb 20. PMID 19234100
- [Result] Kirschenbaum L, Azzi E, Sfeir T, Tietjen P, Astiz M. Effect of continuous lateral rotational therapy on the prevalence of ventilator-associated pneumonia in patients requiring long-term ventilatory care. Crit Care Med. 2002 Sep;30(9):1983-6. doi: 10.1097/00003246-200209000-00006. PMID 12352030
- [Result] Sonnenblick M, Melzer E, Rosin AJ. Body positional effect on gas exchange in unilateral pleural effusion. Chest. 1983 May;83(5):784-6. doi: 10.1378/chest.83.5.784. PMID 6839822
- [Result] Sachdev G, Napolitano LM. Postoperative pulmonary complications: pneumonia and acute respiratory failure. Surg Clin North Am. 2012 Apr;92(2):321-44, ix. doi: 10.1016/j.suc.2012.01.013. PMID 22414416
- [Result] Mirmohammad-Sadeghi M, Etesampour A, Gharipour M, Shariat Z, Nilforoush P, Saeidi M, Mackie M, Sadeghi FM. Early chest tube removal after coronary artery bypass graft surgery. N Am J Med Sci. 2009 Dec;1(7):333-7. doi: 10.4297/najms.2009.7333. PMID 22666720
- [Result] Ahrens T, Kollef M, Stewart J, Shannon W. Effect of kinetic therapy on pulmonary complications. Am J Crit Care. 2004 Sep;13(5):376-83. PMID 15470853
- [Result] Adler J, Malone D. Early mobilization in the intensive care unit: a systematic review. Cardiopulm Phys Ther J. 2012 Mar;23(1):5-13. PMID 22807649
- [Result] Kirkeby-Garstad I, Sellevold OFM, Stenseth R, Skogvoll E, Karevold A. Marked mixed venous desaturation during early mobilization after aortic valve surgery. Anesth Analg. 2004 Feb;98(2):311-317. doi: 10.1213/01.ANE.0000096194.10459.7E. PMID 14742360
- [Result] Kroenke K, Lawrence VA, Theroux JF, Tuley MR. Operative risk in patients with severe obstructive pulmonary disease. Arch Intern Med. 1992 May;152(5):967-71. PMID 1580723